CLINICAL TRIAL: NCT05063812
Title: Performance of a Remote Monitoring Program for Patients Diagnosed With COVID-19
Acronym: RPM
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Neal Sikka, Professor of Emergency Medicine, George Washington University
Other Study IDs: IRB#NCR202520
Record Dates: First submitted 2020-10-01; First posted 2021-10-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Covid19; Infectious Disease; SARS-CoV Infection
Keywords: COVID-19; Emergency Medicine; Remote Patient Monitoring
MeSH Terms: conditions — COVID-19; Communicable Diseases; Severe Acute Respiratory Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — All these patients have been enrolled in the COVID-19 remote patient monitoring program

SUMMARY:
The GW Medical Faculty Associates recently launched a remote monitoring program for patients diagnosed with COVID-19. Patients are provided with a home pulse oximeter and thermometer. Participants complete daily surveys about their symptoms and vital signs and are escalated to receive phone calls and video visits if responses are abnormal.

Investigators would like to complete a study of the program to understand:

1. Operational parameters of program performance, such as how many patients were enrolled and how many patients completed monitoring
2. Clinical course of patients, including their reported symptoms over time and clinical endpoints such as hospitalization or ICU admission
3. Patient satisfaction with program

DETAILED DESCRIPTION:
The SARS-CoV-2 that emerged in late 2019 has been noted to have a wide range of presentations, from asymptomatic and mild cases to those requiring intubation, ECMO, and critical care. As it is a novel pathogen, clinicians and scientists are only beginning understand when and who will require hospital-based resources such as oxygen, hospitalization, or ICU admission. The Medical Faculty Associates (MFA) COVID-19 Remote Monitoring Program (RPM) was developed to provide a daily touchpoint for patients during their COVID-19 course, including ready connection to paramedics and physicians when needed. The program was launched with the goal of identifying clinical decompensation early, maximizing available healthcare capacity, and minimizing nosocomial COVID-19 spread and healthcare worker exposure.

Investigators would like to perform analyses to test multiple hypotheses, including:

1. Patients discharged with a diagnosis of COVID-19 will be able to participate in a remote monitoring program.
2. A COVID-19 remote monitoring program will benefit patients.
3. Patients will be satisfied with their experience of a remote monitoring program and will have lower anxiety about their COVID-19 illness.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed coronavirus infection
* Age >=18
* Primary language English or Spanish

Exclusion Criteria:

* Dementia
* Pregnant > 16 weeks gestation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be all adults enrolled in the COVID-19 Remote Monitoring Program. The investigators anticipate this population to be similar to the GW University Hospital Emergency Department patient population.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient referred | 1 year
  Number of patients referred
Patients enrolled | 1 year
  Number of patients enrolled
Response Rate | 1 year
  Patients giving at least 50% response rate over 10 days
Flagged cases | 1 year
  Number of cases flagged for responses on survey
Telehealth | 1 year
  Number of cases escalated to telehealth
Patient program graduation | 1 year
  Number of patients who graduate from program
Patient unenrollment | 1 year
  Number of patients who unenrolled and for what reason

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University, Department of Emergency Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No